CLINICAL TRIAL: NCT03972423
Title: Impact of a Transmission Checklist in Post Anesthesia Care Unit on Immediate Respiratory Complications
Acronym: TC-IRC
Status: Completed | Type: Observational
Sponsor: Ramsay Générale de Santé (Other)
Collaborators: Dr. Frédéric MARTIN (Unknown)
Responsible Party: Sponsor
Other Study IDs: ID-RCB : 2018-A01825-50
Record Dates: First submitted 2019-05-26; First posted 2019-06-03 (Actual); Last update posted 2020-11-12 (Actual); Status verified 2019-05

CONDITIONS: Anesthesia; Postoperative Complications; Anesthesia Complication
Keywords: checklist; postoperative complication; anesthesia; information transmission; care unit
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- IRCTC group: - The IRCTC group, consisting of all patients included in the 3rd phase of the study and for whom the transmission of information in PACU is carried out using the IRCTC.
  Interventions: Other: With or wiyhout a checklist
- CONTROL group: - The CONTROL group, consisting of all patients included in the 1st phase of the study and for whom the transmission of information in PACU is carried out according to the usual practice.
  Interventions: Other: With or wiyhout a checklist

INTERVENTIONS:
Other: With or wiyhout a checklist — The evaluation of the impact of the use of this Checklist will be done in comparison with the standard transmission practice

SUMMARY:
This work highlighted the beneficial role in terms of carers' satisfaction, quantity and quality of information transmitted.

DETAILED DESCRIPTION:
Communication and information transmission problems are responsible for the majority of serious adverse events. The use of a checklist in the operating theatre has demonstrated its benefit in terms of reducing morbidity and mortality Regarding transmissions between caregivers, numerous studies have shown the great difference between the medical data of a patient in their file and the information transmitted.

The authors recommend using checklists in order to standardise transmissions. This work highlighted the beneficial role in terms of carers' satisfaction, quantity and quality of information transmitted. On the other hand, no study has looked at the reduction of immediate postoperative complications in post anaesthesia care units (PACU).

ELIGIBILITY:
Inclusion Criteria:

* Male or Female over 18 admitted to PACU
* Patient having understood the aims and the methods of the research

  * Patient having expressed their consent to the use of their data.
  * Subject registered with or beneficiary of a social security scheme

Exclusion Criteria:

* Patient participating in another clinical study
* Acute or chronic respiratory insufficiency preoperatively
* Protected patient: adult under guardianship, tutorship or other legal protection, deprived of liberty by judicial or administrative decision
* Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients admitted to PACU
Sampling Method: Non-Probability Sample
Enrollment: 560 (Actual)
Dates: Start 2019-02-18 (Actual); Primary Completion 2019-02-18 (Actual); Study Completion 2020-07-07 (Actual)

PRIMARY OUTCOMES:
arterial oxygen desaturation < 90% | event of at least 15 second duration
  The primary endpoint is defined as the occurrence or not of arterial oxygen desaturation < 90% for more than 15 consecutive seconds in PACU.

CONTACTS AND LOCATIONS:
Overall Officials: Frederic Martin, Principal Investigator — Hospital
Locations (1):
- Les Franciscaines Clinic, Versailles, IDF, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Jaulin F, Lopes T, Martin F. Standardised handover process with checklist improves quality and safety of care in the postanaesthesia care unit: the Postanaesthesia Team Handover trial. Br J Anaesth. 2021 Dec;127(6):962-970. doi: 10.1016/j.bja.2021.07.002. Epub 2021 Aug 5. PMID 34364652